CLINICAL TRIAL: NCT02277691
Title: A Phase 3, Open-label, Multicenter, Long-term Study to Evaluate the Safety and Efficacy of TAK-536, Amlodipine and Hydrochlorothiazide in Subjects With Essential Hypertension
Brief Title: A Phase III Long-term Study of TAK-536TCH in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-536TCH/OCT-001; U1111-1163-0169 (Registry Identifier: WHO); JapicCTI-142689 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Essential Hypertension
Keywords: Pharmacological therapy; Drug Therapy
MeSH Terms: conditions — Essential Hypertension | interventions — Hydrochlorothiazide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-536TCH (Experimental): For 4 weeks during the run-in period, one tablet of TAK-536CCB (as TAK-536/AML, 20 mg/5 mg, respectively) orally, once daily, before or after breakfast.
  For 48 weeks during 52 weeks of the treatment period, one tablet of TAK-536TCH (as TAK-536/AML/HCTZ, 20 mg/5 mg/12.5 mg, respectively) orally, once daily, before or after breakfast. For the remaining 4 weeks of the treatment period, one tablet each of TAK-536CCB and HCTZ 12.5 mg orally, once daily, before or after breakfast.
  Interventions: Drug: TAK-536TCH tablet; Drug: TAK-536CCB tablet; Drug: HCTZ 12.5 mg tablet

INTERVENTIONS:
Drug: TAK-536TCH tablet — TAK-536TCH tablets
Drug: TAK-536CCB tablet — TAK-536CCB tablets
Drug: HCTZ 12.5 mg tablet — HCTZ tablets

SUMMARY:
The purpose of this study is to evaluate the safety of long-term administration of TAK-536, amlodipine (AML), and hydrochlorothiazide (HCTZ) in participants with essential hypertension.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-536TCH. TAK-536TCH is being tested to treat people who have essential hypertension. The study looked at effectiveness and long-term safety of TAK-536TCH in people who took TAK-536CCB in addition to standard care.

The study enrolled 341 patients. Participants received:

* TAK-536CCB (as TAK-536/AML, 20 mg/5 mg) in run-in period,
* TAK-536TCH (as TAK-536/ AML/HCTZ, 20 mg/5 mg/12.5 mg) in treatment period
* TAK-536CCB and HCTZ 12.5 mg in treatment period

All participants were asked to take tablets at the same time each day throughout the study.

This multi-center trial was conducted in Japan. The overall time to participate in this study was 56 weeks (4 weeks run-in period and 52 weeks treatment period). Participants made multiple visits to the clinic during the study.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written informed consent form prior to the initiation of any study procedures.
3. The participant has essential hypertension.
4. The participant has an office sitting systolic blood pressure (SBP) of <180 mmHg and office sitting diastolic blood pressure (DBP) of < 110 mmHg at the start of the run-in period (Week -4). Participants receiving combined therapy with a 3-drug antihypertensive within 4 weeks prior to the start of the run-in period is required to have an office sitting SBP of < 160 mmHg and an office sitting DBP of < 100 mmHg.
5. The participant's office sitting blood pressure at Week -2 and at the end of the run-in period (Week 0) need to be either:

   * Participants without concurrent diabetes mellitus or chronic kidney disease (CKD)*: Sitting SBP of ≥ 140 mmHg or sitting DBP of ≥ 90 mmHg
   * Participants with concurrent diabetes mellitus or CKD*: Sitting SBP of ≥ 130 mmHg or sitting DBP of ≥ 80 mmHg.

     * Estimate glomerular filtration rate according to creatinine (eGFRcreat) of <60 mL/min/1.73 m^2, or urinary albumin (spot urine) of ≥30 μg/mL in laboratory tests performed at Week -2 of the run-in period, and diagnosed with CKD by the investigator or subinvestigator.
6. The participant has an office sitting SBP of < 160 mmHg and office sitting DBP of < 100 mmHg at the end of the run-in period (Week 0).
7. The participant is male or female, aged 20 years or older at the time of providing informed consent.
8. The participant is an outpatient.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agree to use routinely adequate contraception from signing of informed consent through 1 month following the end of the study.

Exclusion Criteria:

1. The participant has received any study drugs within 12 weeks prior to the start of the run-in period.
2. The participant has participated in another clinical study or a post-marketing study within 30 days prior to the start of the run-in period.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g. spouse, parent, child, sibling), or may consent under duress.
4. The participant requires taking prohibited concomitant drugs during the study.
5. The participant has a history of hypersensitivity or allergies to TAK-536, AML, HCTZ, any thiazide diuretic or analog, any dihydropyridine drug, or any analog of TAK-536TCH.
6. The participant is judged by the investigator or subinvestigator to be in danger of experiencing an excessive increase in blood pressure when changing or discontinuing premedication.
7. The participant received combination therapy with antihypertensive drugs of the 3 ingredients contained in TAK-536TCH.
8. The participant received combined therapy with antihypertensive drugs, including 4 or more components, within 4 weeks prior to the start of the run-in period.
9. The participant has secondary or malignant hypertension.
10. The participant has a difference of ≥ 20 mmHg between left and right arms in office sitting SBP at the start of the run-in period (Week -4).
11. The participant has apparent white coat hypertension or exhibits a white coat effect.
12. . The participant has a day-night reversed lifestyle, such as those working during the night.
13. The participant has sleep apnea syndrome requiring treatment.
14. The participant has any of the following cardiovascular diseases:

    * Cardiac disease: Myocardial infarction*, coronary arterial revascularization*, severe valvular disorder, atrial fibrillation, any of the following conditions requiring treatment: angina pectoris, congestive heart failure, arrhythmia
    * Cerebrovascular disorders: Cerebral infarction/cerebral hemorrhage*, transient ischemic attack*
    * Vascular disease: Peripheral artery disease with intermittent claudication, artery dissection, aneurysm
    * Advanced hypertensive retinopathy: With bleeding or exudate/papilledema** * Occurring or performed within 24 weeks of the start of the run-in period ** Observed within 24 weeks of the start of the run-in period
15. The participant has a clinically apparent hepatic disorder (e.g., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at Week -2 of the run-in period ≥ 2.5 times the upper limit of normal (ULN).
16. The participant has a clinically severe renal disorder (e.g., eGFRcreat in laboratory tests performed at Week -2 of run-in period < 30 mL/minute/1.73 m^2).
17. The participant's body fluid sodium or potassium level is markedly low* or high*.

    *Based on normal ranges
18. The participant has gout or a history of gout within 24 weeks of the start of the run-in period or has hyperuricemia requiring drug treatment.
19. The participant has uncontrolled diabetes (e.g., HbA1c ≥ 7.4% in laboratory tests performed at Week -2 of the run-in period).
20. The participant has a malignant tumor.
21. If female, the participant is pregnant or lactating or before giving informed consent, intending to become pregnant or donate ova during or within 1 month after participating in the study.
22. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the run-in period.
23. The participant who, in the opinion of the investigator or subinvestigator, is unsuitable for any other reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (38):
- Japan (38):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Itojima-shi, Fukuoka
  - Kouriyama-shi, Fukushima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Tsukuba, Ibaragi
  - Morioka, Iwate
  - Sakaide-shi, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kawasaki-shi, Kanagawa
  - Kyoto, Kyoto
  - Uji-shi, Kyoto
  - Sendai, Miyagi
  - Hirakata-shi, Osaka
  - Osaka, Osaka
  - Takatsuki-shi, Osaka
  - Saitama-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Yaizu-shi, Shizuoka
  - Chiyoda-ku, Tokyo
  - Choufu-shi, Tokyo
  - Kodaira-shi, Tokyo
  - Koutou-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Choufu-shi
  - Kawasaki-shi
  - Koutou-ku
  - Morioka
  - Sakaide-shi
  - Setagaya-ku
  - Shinagawa-ku
  - Shinjuku-ku
  - Tsukuba
  - Uji-shi
  - Yaizu-shi

REFERENCES:
- [Derived] Rakugi H, Shimizu K, Nishiyama Y, Sano Y, Umeda Y. A phase III, open-label, multicenter study to evaluate the safety and efficacy of long-term triple combination therapy with azilsartan, amlodipine, and hydrochlorothiazide in patients with essential hypertension. Blood Press. 2018 Jun;27(3):125-133. doi: 10.1080/08037051.2017.1412797. Epub 2017 Dec 13. PMID 29235365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 31 investigative sites in Japan, from 07 November 2014 to 25 April 2016.
Pre-assignment Details: Participants with diagnosis of essential hypertension were enrolled in 1 treatment group:TAK-536CCB (TAK-536/ AML,20 mg/5 mg) in run-in period (Week -4 to 0).
Groups:
- TAK-536TCH: For 4 weeks during the run-in period, one tablet of TAK-536CCB (as TAK-536/AML, 20 mg/5 mg, respectively) orally, once daily, before or after breakfast.
  For 48 weeks during 52 weeks of the treatment period, one tablet of TAK-536TCH (as TAK-536/AML/HCTZ, 20 mg/5 mg/12.5 mg, respectively) orally, once daily, before or after breakfast. For the remaining 4 weeks of the treatment period, one tablet each of TAK-536CCB and HCTZ 12.5 mg, orally, once daily, before or after breakfast.
Period: Overall Study
Arm/Group | TAK-536TCH
Started | 341
Completed | 295
Not Completed | 46
Not completed — Pretreatment Event/Adverse Event | 33
Not completed — Voluntary Withdrawal | 7
Not completed — Lack of Efficacy | 5
Not completed — Used Other Antihypertensive Drug | 1

BASELINE CHARACTERISTICS:
Population: Randomized set included all randomized participants.
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 244
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 341
Height [Mean (Standard Deviation); unit: cm] | 164.1 (8.51)
Weight [Mean (Standard Deviation); unit: kg] | 70.80 (12.943)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 26.20 (3.883)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 116
  Current Smoker | 84
  Ex-Smoker | 141
History of Alcohol Consumption [Count of Participants; unit: Participants] — Only participants with history of any alcohol consumption are reported.
  Participants | 120
Duration of Hypertension [Mean (Standard Deviation); unit: years] | 9.42 (7.728)
Concurrent Diabetes Mellitus [Count of Participants; unit: Participants] — Only participants with diabetes mellitus as complication are reported.
  Participants | 90
Concurrent Chronic Kidney Disease [Count of Participants; unit: Participants] — Only participants with chronic kidney disease as complication are reported.
  Participants | 65
Office Sitting Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 143.7 (8.23)
Office Sitting Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 86.2 (9.28)
Estimated Glomerular Filtration Rate According To Creatinine (eGFRcreat) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Male: eGFRcreat (mL/min/1.73 m^2)=194×Cr (mg/dL)-1.094×age (years)-0.287 Female: eGFRcreat (mL/min/1.73 m^2)=194×Cr (mg/dL)-1.094×age (years)-0.287×0.739 Cr: serum creatinine
  mL/min/1.73 m^2 | 78.1 (16.73)
Medical History [Count of Participants; unit: Participants] — Only participants with medical history are reported. Participants may also be counted in more than 1 category.
  Participants
    Cerebrovascular Disorder | 13
    Cardiac Disease | 9
    Vascular Disorder | 1
    Hepatic Disorder | 2
    Dyslipidemia | 1
    Other Medical History | 52
Concurrent Medical Conditions [Count of Participants; unit: Participants] — Only participants with medical conditions are reported. Participants may be counted in more than 1 category.
  Participants
    Cerebrovascular Disorder | 2
    Cardiac Disease | 11
    Vascular Disorder | 21
    Hepatic Disorder | 43
    Dyslipidemia | 174
    Other Concurrent Medical Conditions | 292
Medication History (Antihypertensives) [Count of Participants; unit: Participants] — Only participants with medication history are reported. Participants may be counted in more than 1 category. ARB=angiotensin II receptor blocker, ACE=angiotensin converting enzyme, CCB=calcium channel blocker, β-blockers=beta blockers.
  Participants
    ARBs | 310
    ACE Inhibitors | 9
    CCBs | 313
    Diuretics | 66
    β-blockers | 19
    Other Antihypertensives | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Baseline up to Week 52
Population: The safety analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Participants
  TEAEs | 289
  SAEs | 20

2. Primary Outcome: Number of Participants With Markedly Abnormal Vital Signs Values
Description: Vital signs included supine and standing systolic and diastolic blood pressure (SBP and DBP) respectively and office sitting pulse. Vital signs were considered abnormal if they were beyond the values defined in categories.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Participants
  SBP (Supine) (>180mmHg) | 1
  SBP (Standing) (<85mmHg) | 1
  SBP (Standing) (>180mmHg) | 3
  DBP (Supine) (<50mmHg) | 2
  DBP (Standing) (>110mmHg) | 4
  Office, Sitting Pulse (<50bpm) | 10

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE) Related to Body Weight
Description: Reported TEAE is categorized into investigations System Organ Class (SOC) related to body weight.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Participants
  Weight decreased | 2
  Weight increased | 2

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE) Related to Electrocardiogram (ECG)
Description: Reported TEAE is categorized into cardiac disorders and investigations system organ class (SOC) related to ECG.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Participants
  Atrial fibrillation | 3
  Sinus bradycardia | 1
  QRS axis abnormal | 1

5. Primary Outcome: Number of Participants With Markedly Abnormal Clinical Laboratory Tests
Description: The number of participants with any markedly abnormal clinical laboratory test values collected throughout study. RBC = Red blood cells, ALT = alanine aminotransferase, AST = aspartate aminotransferase, GGT = gamma-glutamyl transferase, LLN = lower limit of normal or lower reference limit, ULN = upper limit of normal or upper reference limit. Laboratory vallues were considered abnormal if they were beyond the values defined in categories.
Time Frame: Baseline up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
Participants
  RBC (< 0.8×LLN×10^6cells/μL) | 5
  Hemoglobin (<0.8 × LLN g/dL) | 2
  Hematocrit (<0.8 × LLN Percent) | 2
  ALT (>3 × ULN U/L) | 4
  AST (>3 × ULN U/L) | 4
  Total Bilirubin (>2.0 mg/dL) | 2
  Creatinine (>2.0 mg/dL) | 1
  Blood Urea Nitrogen (>30 mg/dL) | 20
  GGT (>3 × ULN U/L) | 14
  Eosinophils (>2 × ULN×10^3cells/μL) | 4
  Uric Acid (>13.0 mg/dL) | 1
  Total Cholesterol (>300 mg/dL) | 2
  Triglycerides (>2.5 × ULN mg/dL) | 29
  Potassium (<3.0 mEq/L) | 3
  Sodium (<130 mEq/L) | 3

6. Secondary Outcome: Change From Baseline in Office Trough Sitting Clinic Systolic and Diastolic Blood Pressure at Each Visit
Description: The change in office trough SBP and DBP measured at Weeks 12 last observation was carried forward (LOCF) and 52 (LOCF) relative to baseline. Sitting blood pressure was measured at least 3 times. Each measurement session ended once blood pressure was found stable at 2 consecutive measurements. The average of the last 2 measurements of office sitting blood pressure was used.
Time Frame: Baseline (End of Run-in Period, Week 0) and Weeks 12 (LOCF) and 52 (LOCF)
Population: The full analysis set is defined as the participants who received at least 1 dose of the study drug for the treatment period. Here 'n' is number of participants analyzed at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
mmHg
  Change at Week 12 (LOCF), SBP: number analyzed (Participants) | 339
  Change at Week 12 (LOCF), SBP | -14.4 (12.72)
  Change at Week 52 (LOCF), SBP: number analyzed (Participants) | 339
  Change at Week 52 (LOCF), SBP | -13.9 (12.14)
  Change at Week 12 (LOCF), DBP: number analyzed (Participants) | 339
  Change at Week 12 (LOCF), DBP | -8.6 (8.97)
  Change at Week 52 (LOCF), DBP: number analyzed (Participants) | 339
  Change at Week 52 (LOCF), DBP | -8.3 (9.26)
Statistical Analysis 1: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in office trough SBP at Week 12 (LOCF); Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 2: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in office trough SBP at Week 52 (LOCF); Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 3: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in office trough sitting DBP at Week 12 (LOCF); Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 4: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in office trough sitting DBP at Week 52 (LOCF); Test type: Superiority or Other; p < 0.0001, One sample t-test

7. Secondary Outcome: Change From Baseline in Home Sitting Clinic Systolic and Diastolic Blood Pressure at Each Visit
Description: The change in home morning SPB and DBP measured at End of Week 12, End of Treatment (Up to Week 52) relative to baseline.
Time Frame: Baseline (End of Run-in Period, Week 0), End of Week 12 and End of Treatment (Up to Week 52)
Population: The full analysis set is defined as the participants who received at least 1 dose of the study drug for the treatment period. Here 'n' is number of participants analysed at the given time-point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TAK-536TCH
Number analyzed (Participants) | 341
mmHg
  Change at End of Week 12, Morning SBP: number analyzed (Participants) | 331
  Change at End of Week 12, Morning SBP | -13.9 (10.67)
  Change at EOT (Up to Week 52), Morning SBP: number analyzed (Participants) | 318
  Change at EOT (Up to Week 52), Morning SBP | -12.4 (11.75)
  Change at End of Week 12, Morning DBP: number analyzed (Participants) | 331
  Change at End of Week 12, Morning DBP | -7.9 (6.59)
  Change at EOT (Up to Week 52), Morning DBP: number analyzed (Participants) | 318
  Change at EOT (Up to Week 52), Morning DBP | -6.9 (7.23)
Statistical Analysis 1: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in home SBP, morning at End of Week 12; Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 2: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in home SBP, morning at EOT (Up to Week 52); Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 3: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in home DBP, morning at End of Week 12; Test type: Superiority or Other; p < 0.0001, One sample t-test
Statistical Analysis 4: Comparison: TAK-536TCH; P-value has been estimated for change from baseline in home DBP, morning at EOT (Up to Week 52); Test type: Superiority or Other; p < 0.0001, One sample t-test

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-536TCH
Serious Adverse Events (participants affected / at risk) | 20/341
Other Adverse Events (participants affected / at risk) | 195/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-536TCH (N=341)
Angina pectoris (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 2
Acute abdomen (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Cystitis interstitial (Renal and urinary disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-536TCH (N=341)
Nasopharyngitis (Infections and infestations) | 106
Blood uric acid increased (Investigations) | 86
Hyperuricaemia (Metabolism and nutrition disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 18
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18
Eczema (Skin and subcutaneous tissue disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.